CLINICAL TRIAL: NCT01666678
Title: A Bioavailability Study of Naproxen Sodium and Diphenhydramine Hydrochloride Under Fasting Conditions and Naproxen Sodium and Diphenhydramine Hydrochloride Combination Under Fasting and Fed Conditions
Brief Title: Compare Pharmacokinetic (PK) Profiles of Naproxen Sodium, Diphenhydramine Hydrochloride, and Naproxen Sodium and Diphenhydramine Hydrochloride Combination
Acronym: Morpheus PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 16135
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Therapeutic Equivalence
Keywords: Bioequivalence
MeSH Terms: interventions — Naproxen; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: BAY98-7111
- Arm 2 (Active Comparator)
  Interventions: Drug: Naproxen Sodium (Aleve, BAYH6689)
- Arm 3 (Active Comparator)
  Interventions: Drug: Diphenhydramine HCl
- Arm 4 (Experimental)
  Interventions: Drug: BAY98-7111

INTERVENTIONS:
Drug: BAY98-7111 — 2 x Naproxen Sodium 220 mg / Diphenhydramine HCl 25 mg combination under fasting conditions
  Arms: Arm 1
Drug: Naproxen Sodium (Aleve, BAYH6689) — 2 x Naproxen Sodium 220 mg under fasting conditions
  Arms: Arm 2
Drug: Diphenhydramine HCl — 2 x Diphenhydramine HCl 25 mg under fasting conditions
  Arms: Arm 3
Drug: BAY98-7111 — 2 x Naproxen Sodium 220 mg / Diphenhydramine HCl 25 mg combination under fed conditions
  Arms: Arm 4

SUMMARY:
The purpose of the current trial is to evaluate the bioavailability of a single oral dose of naproxen sodium 440 mg and DPH HCL 50 mg under fasting and fed conditions and currently marketed single ingredient products containing naproxen sodium (2 x Aleve® 220 mg tablets) or DPH HCL (2 Allergy Relief x 25 mg tablets) under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Health, ambulatory male and female subjects between 18 to 55 years of age inclusive
* Body Mass Index (BMI) of approximately 18 to 30 kg/m2; and a total body weight >50 kg (110 lbs)
* Results of screening and clinical laboratory tests are within normal range or considered not clinically significant by the Principal Investigator or Sponsor
* Female subjects of childbearing potential must be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives), e.g., oral or patch contraceptives, intrauterine device, Depo-Provera, or a double barrier and have a negative pregnancy test at Screening and Day 0 for each Dosing Period. Female subjects of non childbearing potential must be amenorrheic for at least 2 years or had a hysterectomy and/or bilateral oophorectomy

Exclusion Criteria:

* History of hypersensitivity to aspirin (ASA), naproxen sodium, NSAIDs, acetaminophen, DPH HCL, and similar pharmacological agents or components of the products
* History of hypersensitivity to any of the food products in the standardized breakfast or cannot consume all food/beverage items contained in the standardized breakfast
* Have taken ASA, ASA-containing products, acetaminophen or any other NSAID (OTC or prescription) 7 days prior to dosing or during the Dosing Periods, other than trial treatment
* Use of any over-the-counter or prescription medications (except acceptable forms of birth control) within 10 days prior to dosing or throughout the trial, unless in the opinion of the Investigator, the medication will not interfere with the trial procedures, data integrity, or compromise the safety of the subject
* Recently had (past 30 days) or plan to have surgery, an invasive procedure, tattoos or piercings during the trial or 1-2 weeks after treatment
* Loss of blood in excess of 500 ml within 56 days of the first dose of trial treatment (e.g., donation, plasmapheresis or injury)
* History of gastrointestinal bleeding or perforation, related to previous NSAID therapy or active or history of recurrent peptic ulcer/hemorrhage (two or more distinct episodes of proven ulceration or bleeding)
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic diseases or malignancies
* Smokers or currently consuming any type of tobacco product(s) including any smoking cessation nicotine-containing product (e.g., nicotine patch, nicotine gum)
* Have taken any vitamin or herbal supplement within 7 days prior to dosing or refuse to refrain from use during the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
AUC(0-tn) (area under the measurement versus time curve from time 0 to the last data point) of naproxen sodium | within 30 minutes prior to dosing (baseline) and 10, 20, 30, 45 minutes and 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 24, and 36 hours post dosing
AUC(0-tn) (area under the measurement versus time curve from time 0 to the last data point) of DPH HCL(Diphenhydramine Hydrochloride) | within 30 minutes prior to dosing (baseline) and 10, 20, 30, 45 minutes and 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 24, and 36 hours post dosing
Cmax(Maximum drug concentration) in plasma of naproxen sodium | within 30 minutes prior to dosing (baseline) and 10, 20, 30, 45 minutes and 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 24, and 36 hours post dosing
Cmax(Maximum drug concentration) in plasma of DPH HCL(Diphenhydramine Hydrochloride) | within 30 minutes prior to dosing (baseline) and 10, 20, 30, 45 minutes and 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 24, and 36 hours post dosing

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Hackensack, New Jersey, United States